CLINICAL TRIAL: NCT01921283
Title: Monitored Anesthesia Care With Propofol Plus Remifentanil During Endoscopic Submucosal Dissection: Evaluation of Bispectral Index Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2011-0347
Record Dates: First submitted 2013-05-22; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Early Gastric Cancer
Keywords: propofol, endoscopy, bispectral index
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS group (Experimental): The BIS group (n=90) was monitored for sedation depth using BIS during ESD.
  Interventions: Device: BIS sensor attachment
- No-BIS group (Active Comparator): The no-BIS group (n=90) was monitored by observer's assessment alertness/sedation scale (OAA/S).
  Interventions: Drug: no- BIS sensor attachment

INTERVENTIONS:
Device: BIS sensor attachment — For double blind method, BIS sensors were attached to all patients, but only BIS-group was measured by the value. BIS monitor was pushed back toward the anesthesiologist so that the physician could not see it. 3 L/min of oxygen was delivered by a nasal cannula to all patients throughout the procedure. Blood pressure was recorded every 5 minutes and heart rate, peripheral oxygen saturation were measured continuously. For induction of sedation, propofol 1 mg/Kg and lidocaine 30mg was administered throughout IV line and immediately followed by continuous infusion of propofol 0.04-0.06 mg/Kg/min and remifentanil 0.05 mcg/Kg/min. The evaluation of sedation depth using OAA/S was performed at 1 minute after propofol administration, endoscopy insertion, submucosal inflation by 1:100000 epinephrine with indigocarmine, initial submucosal dissection and when the patient had restlessness or coughing additively.
  Arms: BIS group
Drug: no- BIS sensor attachment
  Arms: No-BIS group

SUMMARY:
There are clinical usefulness issues associated with bispectral index (BIS) for sedation of endoscopic submucosal dissection (ESD). However, the clinical usefulness of BIS for deep sedation is incompletely described. The purpose of this study is to show that BIS-guided sedation is safe and useful clinically and may provide stable sedation status to physicians and patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I to II.

Exclusion Criteria:

* body mass index (BMI) over 35 (Kg/m2)
* hepatic or renal insufficiency
* history of allergy to the drugs used
* history of administration of anxiolytics, narcotics, antipsychotics, opioid.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
procedure satisfaction score of propofol addition | an average time for 1 week from propofol addition
  The evaluation of sedation depth using OAA/S will be performed at 1 minute after propofol administration, endoscopy insertion, submucosal inflation by 1:100000 epinephrine with indigocarmine, initial submucosal dissection and when the patient have restlessness or coughing additively.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Bell JK, Laasch HU, Wilbraham L, England RE, Morris JA, Martin DF. Bispectral index monitoring for conscious sedation in intervention: better, safer, faster. Clin Radiol. 2004 Dec;59(12):1106-13. doi: 10.1016/j.crad.2004.04.008. PMID 15556593
- [Background] Sugimoto T, Okamoto M, Mitsuno Y, Kondo S, Ogura K, Ohmae T, Mizuno H, Yoshida S, Isomura Y, Yamaji Y, Kawabe T, Omata M, Koike K. Endoscopic submucosal dissection is an effective and safe therapy for early gastric neoplasms: a multicenter feasible study. J Clin Gastroenterol. 2012 Feb;46(2):124-9. doi: 10.1097/MCG.0b013e31822f3988. PMID 21959325
- [Background] Kim SG. Endoscopic treatment for early gastric cancer. J Gastric Cancer. 2011 Sep;11(3):146-54. doi: 10.5230/jgc.2011.11.3.146. Epub 2011 Sep 29. PMID 22076219
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- [Background] Cohen LB, Delegge MH, Aisenberg J, Brill JV, Inadomi JM, Kochman ML, Piorkowski JD Jr; AGA Institute. AGA Institute review of endoscopic sedation. Gastroenterology. 2007 Aug;133(2):675-701. doi: 10.1053/j.gastro.2007.06.002. No abstract available. PMID 17681185
- [Background] Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy; Lichtenstein DR, Jagannath S, Baron TH, Anderson MA, Banerjee S, Dominitz JA, Fanelli RD, Gan SI, Harrison ME, Ikenberry SO, Shen B, Stewart L, Khan K, Vargo JJ. Sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2008 Nov;68(5):815-26. doi: 10.1016/j.gie.2008.09.029. No abstract available. PMID 18984096
- [Background] Imagawa A, Fujiki S, Kawahara Y, Matsushita H, Ota S, Tomoda T, Morito Y, Sakakihara I, Fujimoto T, Taira A, Tsugeno H, Kawano S, Yagi S, Takenaka R. Satisfaction with bispectral index monitoring of propofol-mediated sedation during endoscopic submucosal dissection: a prospective, randomized study. Endoscopy. 2008 Nov;40(11):905-9. doi: 10.1055/s-2008-1077641. PMID 19023932
- [Background] Kang KJ, Min BH, Lee MJ, Lim HS, Kim JY, Lee JH, Chang DK, Kim YH, Rhee PL, Rhee JC, Kim JJ. Efficacy of Bispectral Index Monitoring for Midazolam and Meperidine Induced Sedation during Endoscopic Submucosal Dissection: A Prospective, Randomized Controlled Study. Gut Liver. 2011 Jun;5(2):160-4. doi: 10.5009/gnl.2011.5.2.160. Epub 2011 Jun 24. PMID 21814595